CLINICAL TRIAL: NCT04776434
Title: SUCCESS (SelUtion, Safety, effiCaCy, hEalth economicS and promS) PTA Study
Acronym: SUCCESS PTA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.A. Med Alliance S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2020-01
Record Dates: First submitted 2021-02-10; First posted 2021-03-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SELUTION SLR™ DEB (Experimental): Med Alliance SELUTION SLR™ 018 DEB Sirolimus Eluting Balloon Catheter.
  Interventions: Device: SELUTION SLR™ (Sustained Limus Release) drug eluting balloon (DEB)

INTERVENTIONS:
Device: SELUTION SLR™ (Sustained Limus Release) drug eluting balloon (DEB) — This study will capture data from the use of the SELUTION SLR according to its approved labelling.

SUMMARY:
Open label, real-world, prospective, multi-center, single arm, post-market surveillance study of the SELUTION SLR™ (Sustained Limus Release) drug eluting balloon (DEB).

DETAILED DESCRIPTION:
Open label, real-world, prospective, multi-center, single arm, post-market surveillance study of the SELUTION SLR™ (Sustained Limus Release) drug eluting balloon (DEB).

This study will capture data from the use of the SELUTION SLR according to its approved labelling. Each indication for use will have a specific data sets in addition to generic data sets that are common across all indications.

Patients will be followed for 5 years post-procedure to obtain safety and efficacy data. A health economic analysis will be made comparing data between countries within the study and to published data for existing treatment options. Generic and disease specific Patient Reported Outcome Measures (PROMs) will be used to measure the impact of the intervention on the overall health status of patients.

Imaging data collection for patients whose standard of care includes imaging follow-up will be captured and analysed.

Data will be collected from any subject who receives a CE marked device for treatment of a peripheral (i.e. non-cardiovascular) vascular lesion.

Data analysis will be stratified by lesion location.

ELIGIBILITY:
Inclusion Criteria:

* Subject age is ≥ 18 years
* Subject is able and willing to provide informed consent
* Subject is suitable for treatment with a MedAlliance SELUTION SLR DEB according to the current Instruction for use.

Exclusion Criteria:

* In the opinion of the treating investigator the subject has a life expectancy of less than 12 months
* In the opinion of the treating investigator the subject is unlikely to comply with the study follow-up regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinically Driven Target Lesion Revascularization | 1 year after treatment
  The primary endpoint will be freedom from Clinically Driven Target Lesion Revascularisation (CD-TLR) at 1-year post-intervention.

SECONDARY OUTCOMES:
Device Success | At end of procedure
  Successful delivery, balloon inflation, deflation and retrieval of the intact study device without burst below rated burst pressure.
Procedure success | At end of procedure
  Device success and residual stenosis ≤50% at the end of the procedure.
Clinical success | At discharge after procedure
  Procedural success without procedural complications (death, major target limb amputation, thrombosis of the target lesion or TLR) prior to discharge.
Major Adverse Limb Events (MALE) composite endpoint | At discharge after procedure and 1, 6, 12, 24, 36, 48 and 60 months
  Severe limb ischemia leading to an intervention or major vascular amputation (above the ankle).
Major Cardiac Events Major Cardiac Events | At 1, 6, 12, 24, 36,48, 60 months
  MI, Stroke, Cardiovascular death
Death | At 1, 6, 12, 24, 36, 48, 60 months
  All-cause, cardiac, device related, procedure related
TLR | At 1, 6, 12, 24, 36, 48, 60 months
  Number of Target Lesion Revascularizations
TVR | At 1, 6, 12, 24, 36, 48, 60 months
  Number of Target Vessel Revascularizations
Time to first CD-TLR | up to 60 months
  Time to first Clinically Driven Target Lesion Revascularization
Target limb revascularization | At 1, 6, 12, 24, 36, 48, 60 months
  Number of Target limb revascularizations
Thrombosis at the target site | At 1 month
  Number of Thrombosis at the target site
Amputation | up to 60 months
  Number of Amputations
Rutherford Classification score | At 6, 12, 24, 36, 48, 60 months
  Change in Rutherford Classification score from baseline (Scale from 0 to 6, higher score means worse outcome.
Ankle Brachial Index (ABI) | At 6, 12 months only
  Change in ankle brachial index (ABI) from baseline
Pedal pulse | 6, 12 months only
  Presence of Pedal pulse
Wound status if applicable | 6, 12 months only
  location, size, infection, status, Wound, Ischemia and Foot Infection (WIfI) classification system score
Kawarada Classification score | At end of procedure
  Change from baseline to end of procedure to assess change in severity of Pedal Artery Disease

CONTACTS AND LOCATIONS:
Locations (27):
- Hospital Italiano La Plata, La Plata, Argentina
- Germany (12):
  - Klinikum Hochsauerland, Arnsberg
  - Universitätsklinikum Freiburg, Bad Krozingen
  - Krankenhaus Buchholz, Buchholz
  - Universitätsklinikum Essen, Essen
  - DIAKO Krankenhaus, Flensburg
  - Medizinisches Versorgungszentrum, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - SRH Klinikum Karlsbad - Langensteinbach, Langensteinbach
  - LMU Klinikum Campus Großhadern, München
  - Universitätsklinikum Tübingen, Tübingen
  - Grn Klinik Weinheim, Weinheim
  - Universitätsklinikum Würzburg, Würzburg
- Greece (3):
  - Athens Medical Center, Athens
  - Attikon University Hospital, Athens
  - General University Hospital of Patras, Pátrai
- Elisabeth - TweeSteden Ziekenhuis, Tilburg, Netherlands
- National University Hospital Singapore (NUHS), Singapore, Singapore
- Trnava University Hospital, Trnava, Slovakia
- Switzerland (3):
  - Kantonsspital Aarau, Aarau
  - Hôpitaux Universitaires de Genève (HUG), Geneva
  - Luzerner Kantonsspital, Lucerne
- United Kingdom (5):
  - Frimley Park Hospital, Frimley
  - University Hospitals of Leicester NHS Trust, Leicester
  - Barts Health NHS Trust (ROYAL HOSPITAL LONDON), London
  - Guy's & St Thomas Hospital, London
  - East Surrey Hospital, Redhill

IPD SHARING:
Plan to Share IPD: Undecided